CLINICAL TRIAL: NCT02983786
Title: Detection of Cerebral Ischemia With a Noninvasive Neurometabolic Optical Monitor
Acronym: NNOM
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 819681
Record Dates: First submitted 2015-12-03; First posted 2016-12-06 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Traumatic Brain Injury; Ischemic Stroke; Intracerebral Hemorrhage; Subarachnoid Hemorrhage; Acute Anoxic Encephalopathy
MeSH Terms: conditions — Brain Injuries, Traumatic; Ischemic Stroke; Cerebral Hemorrhage; Subarachnoid Hemorrhage | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Non-Invasive Monitoring: One non-invasive optode patch will be placed adjacent to the area of invasive monitoring and the second patch will be placed contralaterally. (12 hrs. daily is chosen primarily for budgetary reasons). The information for the non-invasive technology will be compared to the invasive technology.
  ICG (Indocyanine Green) will be injected to derive absolute CBF and calibrate the DCS monitor to yield continuous absolute CBF. During each 12-hour monitoring session, for up to 14 days, the ICG will be injected at baseline(0.2 mg/kg,(4), every four hours (or less if signal is stable).
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — ICG will be injected to derive absolute CBF and calibrate the DCS monitor to yield continuous absolute CBF. During each 12-hour monitoring session, for up to 14 days, the ICG will be injected at baseline(0.2 mg/kg,(4), every four hours (or less if signal is stable).
  Other Names: Indocyanine Green Injection

SUMMARY:
The goals of the project are to evaluate a noninvasive monitor of brain metabolism and blood flow in critically ill humans. If validated, such a reliable noninvasive brain blood flow and metabolism monitor, by allowing physiologic and pharmacologic decisions based on real-time brain physiology, potentially will become an important tool for clinicians in their efforts to prevent additional brain tissue death in patients admitted with stroke, brain hemorrhage and traumatic brain injury.

DETAILED DESCRIPTION:
Many critically ill patients are admitted to the hospital with no infarcted brain tissue and yet, after a period of extremely intense and expensive critical care, the patients are discharged with new hospital-acquired dead brain tissue, with associated life-long disability or brain death. This situation arises from the critical barrier of there being no straightforward bedside methods to monitor cerebral blood flow (CBF) and its adequacy during progression of post-insult secondary brain damage. This is important because of the expectation that decrements in CBF in dangerous excess of decrements in cerebral metabolic rate for oxygen (CMRO2), if detected early, can be treated to avert brain infarction. Clinical examples of this issue, among many others, include post ischemic stroke edema, post thrombolysis hyperemia or occlusion, post SAH vasospasm, hyperemic and oligemic intracranial hypertension after traumatic brain injury or stroke, ICH associated global ischemia, and intra and post carotid endarterectomy oligemia and hyperperfusion.

Critical care physicians need a bedside monitor of CBF coupled to CMRO2. The CMRO2 data will allow delineation of adequacy of CBF as occasionally CBF decrements are simply matching changes in CMRO2. The lack of such monitoring capability has resulted in clinicians making often not helpful therapeutic decisions directed to non-neurologic endpoints, e.g., blood pressure, PaCO2 and so on, "hoping" that such interventions will have a desired effect on brain perfusion and metabolism.

Diffuse Correlation Spectroscopy (DCS) and Diffuse Optical Spectroscopy (DOS) are promising NNOM optical techniques under development at UPenn (Dr. Arjun Yodh) which can provide continuous bedside quantitative CBF, CMRO2 and oxygen extraction fraction (OEF) information. Determination of capability to detect anaerobic conditions, as the investigators propose doing, will make feasible the notion of individualized CBF, CMRO2, and OEF measurement and brain-directed therapeutic optimization by bedside caregivers. This will eventually support a significant change in the way Neurocritical Care is practiced, titrating therapy to neurophysiologic rather than cardiovascular/ pulmonary endpoints. UPenn research techniques presently provide information on relative quantitative changes in CBF and CMRO2 from baseline. The investigators propose also developing a method for measurement of absolute CBF and CMRO2 and further validating the absolute CBF against invasive thermodilution (ThD) CBF techniques. The investigators' long range goal and overall objective is to prevent in-hospital brain tissue death through development of improved bedside CBF/ CMRO2/OEF (NNOM) monitoring techniques.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be age greater than or equal to 18 years, the diagnosis of SAH, TBI, ICH, and/or (PIAE) after cardiac arrest (post cardiac arrest coma) with GCS less than or equal to 8, endotracheal intubation, clinical indications for invasive Neuromonitoring, and family/guardian informed consent.

Exclusion Criteria:

1. coagulation or platelet problems which cannot be corrected based on clinical indications
2. anatomic abnormalities in skull or brain tissue precluding appropriate placement of an invasive brain monitor
3. ongoing CNS or scalp infection,
4. allergy to indocyanine green dye
5. pregnancy
6. lactation or pumping breast milk for the purpose of feeding an infant
7. increased bilirubin suggestive of cholestasis or biliary obstruction, (8) allergy to iodide

(9) severity of injury which leads the team or family to conclude that further advance medical care would be futile and limitation of the level of support is requested.

Woman of childbearing potential will be excluded by urine or serum pregnancy test prior to conducting any study related procedures. . There is not a risk of pregnancy during this study as comatose patients will be monitored 24 hours a day in Intensive Care Units which have full visibility of patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria will be age greater than or equal to 18 years, the diagnosis of SAH, TBI, ICH, and/or PIAE after cardiac arrest (post cardiac arrest coma) with GCS less than or equal to 8 (coma- clinical indications for invasive neuromonitoring), endotracheal intubation, clinical indications for invasive neuromonitoring, and family/guardian informed consent.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-12; Primary Completion 2018-10 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
The outcome variable will be the degree of correlation of ThD (thermodilution) CBF with optical CBF (cerebral blood flow). | 12 days
  Determine if the optical monitoring device's assessment of CBF is valid.

SECONDARY OUTCOMES:
The outcome variable will be whether the optical monitoring system detects an anaerobic condition based on specific criteria of low ThD CBF, low brain PO2(PbrO2), and high microdialysis lactate pyruvate ratio ( LPR). | 12 Days
  Determine if the optical monitoring system can detect an anaerobic adverse condition in the brain which might lead to neural injury.

OTHER OUTCOMES:
The outcome variable will be a determination of characteristics of trends in systemic and neurophysiologic data which predict the later development of an anaerobic condition in the brain. | 12 days
  Predict the later onset of a brain anaerobic condition.

CONTACTS AND LOCATIONS:
Overall Officials: W. Andrew Kofke, MD, Principal Investigator — University of Pennsylvania Health System
Locations (1):
- University of Pennylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No, study data only remains with the study team. update reports will be submitted to the NIH, however individual patient data will not be included.